CLINICAL TRIAL: NCT04987723
Title: A Mechanistic Exploratory Study of AF-induced Cardiac Dysfunction and Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 272775
Record Dates: First submitted 2021-07-14; First posted 2021-08-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: atrial fibrillation; heart failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AF + HFrEF cohort (Other): Left Ventricular Ejection Fraction (LVEF) < 50% by echocardiogram during routine screening or within 12 months prior to enrolment day. The echo must have been performed >3 weeks after optimisation of HF and rate control therapies, otherwise repeat imaging will be performed after this has been achieved
  With
  NYHA functional status II-III at the enrolment visit.
  Interventions: Other: Holter monitoring; Other: stress echocardiography; Other: Cardiac MRI; Other: Patient questionnaires
- AF + symptoms cohort (Other): Left Ventricular Ejection Fraction (LVEF) > 50% by echocardiogram during routine screening or within 12 months prior to enrolment day
  With
  modified European Heart Rhythm Association symptom classification 2b-4.
  Interventions: Other: Holter monitoring; Other: Patient questionnaires

INTERVENTIONS:
Other: Holter monitoring — Assessment of HRV shall be performed in all enrolled patients. Ventricular HRV will be derived from a continuous 24-hour period of a 48-hour ambulatory Holter recording during AF. Participants will be requested to avoid alcohol and caffeine from 24-hours prior to fitting and any activity more strenuous than walking for the recording duration. After initial fitting, a 20-minute high-resolution ECG recording will be performed lying supine at rest.
  Other Names: Heart rate variability recording
Other: stress echocardiography — Echocardiography will be performed using a GE Vivid 9 echocardiography machine (Vingmed-General Electric, Horten, Norway) equipped with a phased-array 3.5 MHz transducer. All measurements will be made according to the guidelines set by the British Society of Echocardiography.
  Other Names: assessment of cardiac reserve
  Arms: AF + HFrEF cohort
Other: Cardiac MRI — Contraindications to MRI will be excluded using the appropriate departmental screening forms. A trained scanner operator or radiographer will co-ordinate and supervise the scan. Cardiac MRI will be performed at 1.5T (Aera, Siemens Healthineers, Erlangen, Germany) with a protocol consisting of cine imaging, stress and rest perfusion, and late gadolinium enhancement (LGE).
  Arms: AF + HFrEF cohort
Other: Patient questionnaires — Two validated Health Related Quality of Life (HRQoL) surveys designed for patients with AF will be used; the AF Effect on Quality of Life (AFEQT) and Barts AF Patient reported objective measure (PROM).
  Other Names: AFeQT questionnaire and the Barts AF PROM questionnaire

SUMMARY:
Although the heart rhythm disorder Atrial Fibrillation (AF) affects 2% of the population, the impact it has on an effected individual can be highly variable. Some people are asymptomatic whilst others can experience debilitating symptoms or heart failure (HF)- weakness of the heart muscle. The reason why this variability exists in unknown and how AF actually drives HF is unclear. HF can also be caused by many other reasons and it can be difficult to identify those patients with HF caused by AF versus patients with AF but their HF is due to a different reason. This is important as it would help us to identify those patients most likely to improve their heart function after the treatment of AF and thus gain more from invasive treatments like AF catheter ablation; which is effective at restoring normal heart rhythm but has some risks attached.

The investigators suspect the characteristics of the AF, such as how irregularly it makes the heartbeat, can be used to predict who will respond better. Studies of heart cells in the lab as well as animal models have suggested this characteristic may be the cause of AF-induced heart muscle weakness and reduce cardiac output, making it a potential predictor that can be measured. Other potential predictors will be measured during pre-procedural scans and tests too. The investigators will also explore whether there are predictors of which patients gain the most symptomatic benefit and gain insight into why some people develop symptoms of AF, whereas others do not.

By studying the structural and functional sequelae of catheter ablation in patients with HF the investigators hope to better understand the relationship between the two diseases.

ELIGIBILITY:
Inclusion Criteria:

* Referred for first AFCA procedure by their responsible physician.
* Persistent AF captured on ECG but not in continuous AF for more than 3 years. (Persistent AF will be defined as any continuous episode lasting longer than 7 days or requiring intervention to restore sinus rhythm after this time.)
* Participants must have either:

  * Left Ventricular Ejection Fraction (LVEF) < 50% by echocardiogram during routine screening or within 12 months prior to enrolment day. The echo must have been performed >3 weeks after optimisation of HF and rate control therapies, otherwise repeat imaging will be performed after this has been achieved

With:

o NYHA functional status II-III at the enrolment visit.

Or:

o Left Ventricular Ejection Fraction (LVEF) >50% by echocardiogram during routine screening or within 12 months prior to enrolment day.

With:

o modified European Heart Rhythm Association 2a-4.

Exclusion Criteria:

* Previous left atrial ablation procedure or surgery.
* Contraindication to chronic anticoagulation therapy or heparin
* Unable or unwilling to consent to investigation and follow-up requirements or inability to comply with planned study procedures.
* LA anteroposterior diameter ≥ 5.5 cm or indexed LA volume ≥ 50mL/m2 on echo.
* Recent (last 6 months) event that may impact LV function- myocardial infarction, coronary revascularization, pacemaker or cardiac resynchronization therapy.
* AF suspected to be due to a reversible cause (e.g. hyperthyroidism, recent surgery)
* Acute coronary syndrome within 4 weeks as defined by ECG ST segment depression or prominent T-wave inversion and/or positive biomarkers of necrosis (e.g. troponin) in the absence of ST-segment elevation and in an appropriate clinical setting (chest discomfort or angina equivalent).
* Cardiac surgery, angioplasty, or cerebrovascular accident within 4 weeks prior to enrolment.
* Life expectancy less than 1 year.
* Chronic kidney disease stage 4 or 5.
* Any of the below cardiac diagnoses:

  * Hypertrophic obstructive cardiomyopathy
  * Severe valvular disease
  * Restrictive or constrictive cardiomyopathy, including known amyloidosis, sarcoidosis,
  * haemochromatosis
  * Complex congenital heart disease
  * Constrictive pericarditis
  * Severe pulmonary hypertension (RVSP > 60 mmHg),
  * Non-cardiac pulmonary oedema
  * Active myocarditis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Correlation co-efficient of HRV measures with change in cardiac function | 6 months after catheter ablation
  This will be calculated in the AF + HFreF arm
  Cardiac function will be measured as three endpoints:
  * LVEF on echocardiography
  * Serum NT-proBNP
  * VO2 peak on CPET

SECONDARY OUTCOMES:
Correlation co-efficient of LA strain with change in cardiac function | 6 months after catheter ablation
  This will be calculated in the AF + HFreF arm
  Cardiac function will be measured as three endpoints:
  * LVEF on echocardiography
  * Serum NT-proBNP
  * VO2 peak on CPET
Correlation co-efficient of HRV measures with change in score on validated AF PROM questionnaire | 6 months
  This will be calculated for each study arm independently. The scores from the
  * AFeQT survey
  * Barts AF PROM survey will be used

OTHER OUTCOMES:
Relative frequency of pre-specified genetic variants in participants retrospectively deemed to have AF-induced HF as compared to a reference cohort. | 1 day [At baseline assessment]
Correlation co-efficient between R-R intervals derived from single-lead ECG time-series from the selected devices whilst recording simultaneously. | 1 day [At baseline assessment]
  Correlation co-efficient (r) between HRV measured using gold standard ECG monitoring and wearable-derived HRV.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunter RJ, Berriman TJ, Diab I, Kamdar R, Richmond L, Baker V, Goromonzi F, Sawhney V, Duncan E, Page SP, Ullah W, Unsworth B, Mayet J, Dhinoja M, Earley MJ, Sporton S, Schilling RJ. A randomized controlled trial of catheter ablation versus medical treatment of atrial fibrillation in heart failure (the CAMTAF trial). Circ Arrhythm Electrophysiol. 2014 Feb;7(1):31-8. doi: 10.1161/CIRCEP.113.000806. Epub 2014 Jan 1. PMID 24382410
- [Derived] Ahluwalia N, Honarbakhsh S, Abbass H, Joshi A, Chow AWC, Dhinoja M, Petersen SE, Hunter RJ, Lloyd G, Schilling RJ. Characterisation of patients who develop atrial fibrillation-induced cardiomyopathy. Open Heart. 2024 Nov 27;11(2):e002955. doi: 10.1136/openhrt-2024-002955. PMID 39608861